CLINICAL TRIAL: NCT04108000
Title: SPIRIT for Persons With Dementia and Complex Multimorbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mi-Kyung Song, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00094859a; 3R01NR017018 (NIH); 5R01AG057714 (NIH)
Record Dates: First submitted 2019-09-26; First posted 2019-09-27 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: End Stage Renal Disease
Keywords: Dementia; Nursing; Nephrology; Behavioral research; Social research
MeSH Terms: conditions — Kidney Failure, Chronic; Dementia

STUDY DESIGN:
Intervention Model Description: 30 pairs of patients and their caregivers (surrogates) will be randomized to either receive the SPIRIT intervention or standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPIRIT-Dementia (Experimental): Patients and their surrogates randomized to this study arm will receive the SPIRIT-dementia intervention.
  Interventions: Behavioral: SPIRIT-Dementia
- Usual Care (Active Comparator): Patients and surrogates randomized to this study arm will receive the standard information about advance directives that is provided at the time of diagnosis.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: SPIRIT-Dementia — The interventionist will begin the SPIRIT-dementia session by assessing the patient's and surrogate's cognitive, emotional, and spiritual/religious representations of the patient's illness, prognosis, and end-of-life care. Individualized information will be provided about the effectiveness of life-sustaining treatment for people with end-organ failure, and the patient will examine their values about life-sustaining treatment at the end of life. The interventionist will help the surrogate prepare for end-of-life decision-making and for the emotional burden of decision-making. A Goals-of-Care document will be completed at the end of the session. The delivery of SPIRIT-dementia incorporates "enhanced consent techniques," such as reducing information load by proceeding in manageable segments, offering repetition of material, opportunity for rehearsal, and using targeted questioning to verify adequate comprehension prior to eliciting preferences for goals of care.
  Arms: SPIRIT-Dementia
Behavioral: Usual Care — As required by Centers for Medicare and Medicaid Services (CMS) written information on advance directives is provided to a patient on the first day of dialysis, and a social worker reviews this information with patients and encourages them to complete an advance directive.
  Arms: Usual Care

SUMMARY:
In this study, 30 patient and caregiver dyads will be randomized to receive the SPIRIT-dementia intervention or usual care. Participants will be follow-up with 2-3 days after the intervention to evaluate the impact of SPIRIT on preparedness outcomes. Additional follow up with caregivers will occur 6 months later.

DETAILED DESCRIPTION:
Cognitive impairment or dementia, usually vascular dementia or Alzheimer's, co-occur in approximately 38% of patients with end stage renal disease (ESRD). When dementia is superimposed on ESRD, the risk for poor outcomes, including disability, hospitalization and death, sharply increases. Similarly, initiating dialysis in older adults with multiple comorbidities, including dementia, does not offer survival benefit. However, advance care planning (ACP) discussions with dialysis patients rarely occur. The reality of ESRD plus dementia is that most of these patients are likely to die or progress to advanced dementia without ever engaging in ACP discussions before the cognitive window of opportunity closes. Moreover, persons with dementia (regardless of their cognitive impairment level) are routinely excluded from clinical trials of ACP, largely because investigators assume that these people do not have the cognitive capability to appreciate the complexity of ACP. In an on-going study ("SPIRIT in Dementia") the researchers carefully adapted SPIRIT for persons with mild to moderate dementia (mostly due to Alzheimer's) and their surrogates. In a sample of 23 dementia patients without complex multimorbidity and their surrogates, the researchers were able to conclude that meaningful ACP conversations were possible even for individuals with moderate dementia. Based on these findings, this supplement study will leverage the infrastructure of the parent SPIRIT in ESRD trial to pilot test the adapted SPIRIT intervention for patients with ESRD plus dementia as a model for determining whether patients with dementia superimposed on complex multimorbidity can fully participate in ACP discussion.

This purpose of this pilot randomized controlled trial with 30 patient and caregiver dyads is to:

* estimate the effects of the SPIRIT-dementia intervention on: (a) preparedness outcomes for end-of-life decision making (defined as dyad congruence on goals of care, patient decisional conflict, and surrogate decision-making confidence) 2-3 days post-intervention, and (b) care decisions (withdrawal from dialysis, Do-Not-Resuscitate order, hospice enrollment) assessed at 6 months post-intervention, or the patient's death, whichever occurs first,
* estimate the effects of the SPIRIT-dementia intervention on surrogates' post-bereavement distress (anxiety and depression symptoms) at 1 month after the patient's death, and
* explore the relationships among patients' cognitive status, decision-making capacity and their ability to express end-of-life wishes.

ELIGIBILITY:
Patient Inclusion Criteria:

* receiving in-center hemodialysis
* diagnosed with dementia or having mild to moderate cognitive impairment based on a Montreal Cognitive Assessment (MoCA) score 13-25 or a Saint Louis University Mental Status (SLUMS) score < 27 (high school education) or < 25 (less than high school education)
* able to understand and speak English
* a University of California San Diego Brief Assessment of Capacity to Consent (UBACC) score of 11 or higher

Exclusion Criteria:

* lack of an available surrogate
* uncompensated hearing deficits
* already enrolled in hospice

Surrogate Inclusion Criteria:

* 18 years or older
* be chosen by the patient
* able to understand and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Kyung Song, RN, PhD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory Dialysis at Northside, Atlanta, Georgia
  - Emory Dialysis at Greenbriar, Atlanta, Georgia
  - Emory Dialysis at North Decatur, Decatur, Georgia
  - Emory Dialysis at Candler, Decatur, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from multiple dialysis centers in Georgia, USA. Participant enrollment began on February 14, 2020, and follow-up assessments for the primary outcome measures were completed on March 24, 2023.
Pre-assignment Details: Research team chose individual randomization because intervention spillover to the control condition was very unlikely. Race was used (white vs non-white) as stratification factor to ensure equal allocation of race to each condition to control for race as a confounder. Intervention was delivered by a trained interventionist, in person, or virtually due to COVID-19, and thus it was nearly impossible for care providers to obtain the knowledge and skill related to SPIRIT to change their practice.
Groups:
- SPIRIT-Dementia -Patients: Patients and their surrogates randomized to this study arm will receive the SPIRIT-dementia intervention.
  SPIRIT-Dementia: The interventionist will begin the SPIRIT-dementia session by assessing the patient's and surrogate's cognitive, emotional, and spiritual/religious representations of the patient's illness, prognosis, and end-of-life care. Individualized information will be provided about the effectiveness of life-sustaining treatment for people with end-organ failure, and the patient will examine their values about life-sustaining treatment at the end of life. The interventionist will help the surrogate prepare for end-of-life decision-making and for the emotional burden of decision-making. A Goals-of-Care document will be completed at the end of the session. The delivery of SPIRIT-dementia incorporates "enhanced consent techniques," such as reducing information load by proceeding in manageable segments, offering repetition of material, an opportunity for rehearsal, and using targeted questioning to verify adequate comprehension prior to eliciting preferences for goals of care.
- SPIRIT-Dementia -Surrogate: Surrogates of patients randomized to this study arm will receive the SPIRIT-dementia intervention.
  SPIRIT-Dementia: The interventionist will begin the SPIRIT-dementia session by assessing the patient's and surrogate's cognitive, emotional, and spiritual/religious representations of the patient's illness, prognosis, and end-of-life care. Individualized information will be provided about the effectiveness of life-sustaining treatment for people with end-organ failure, and the patient will examine their values about life-sustaining treatment at the end of life. The interventionist will help the surrogate prepare for end-of-life decision-making and for the emotional burden of decision-making. A Goals-of-Care document will be completed at the end of the session. The delivery of SPIRIT-dementia incorporates "enhanced consent techniques," such as reducing information load by proceeding in manageable segments, offering repetition of material, an opportunity for rehearsal, and using targeted questioning to verify adequate comprehension prior to eliciting preferences for goals of care.
- Usual Care - Patients: Patients and surrogates randomized to this study arm will receive the standard information about advance directives that are provided at the time of diagnosis.
  Usual Care: As required by the Centers for Medicare and Medicaid Services (CMS) written information on advance directives is provided to a patient on the first day of dialysis, and a social worker reviews this information with patients and encourages them to complete an advance directive.
- Usual Care - Surrogates: Surrogates of patients randomized to this study arm will receive the standard information about advance directives that are provided at the time of diagnosis.
  Usual Care: As required by the Centers for Medicare and Medicaid Services (CMS) written information on advance directives is provided to a patient on the first day of dialysis, and a social worker reviews this information with patients and encourages them to complete an advance directive.
Period: Overall Study
Arm/Group | SPIRIT-Dementia -Patients | SPIRIT-Dementia -Surrogate | Usual Care - Patients | Usual Care - Surrogates
Started | 9 | 9 | 10 | 10
Completed | 6 | 6 | 9 | 9
Not Completed | 3 | 3 | 1 | 1
Not completed — Death of patient | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0
Not completed — Death of surrogate partner | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPIRIT-Dementia -Patients | SPIRIT-Dementia -Surrogate | Usual Care - Patients | Usual Care - Surrogates | Total
Number analyzed (Participants) | 9 | 9 | 10 | 10 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.44 (8.35) | 57.56 (11.41) | 63.40 (11.43) | 53.20 (12.19) | 58.42 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 4 | 5 | 23
  Male | 3 | 1 | 6 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 9 | 9 | 8 | 9 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 9 | 8 | 8 | 34
  White | 0 | 0 | 2 | 2 | 4
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 10 | 10 | 38

OUTCOME MEASURES:

1. Primary Outcome: Dyad Congruence
Description: Dyad congruence will be assessed using the Goals-of-Care Tool which includes two scenarios describing medical conditions commonly occurring in ESRD patients. Possible responses to the scenarios are: "The goals of care should focus on delaying my death, and thus I want to continue life-sustaining treatment", "The goals of care should focus on my comfort and peace, and thus I do not want life-sustaining treatment, including dialysis", and "I am not sure". Patients and surrogates complete this tool independently and their responses are then compared to determine dyad congruence.
Time Frame: Baseline, 2 Days Post-intervention
Population: The Unit of measure and analysis is a dyad (patient-surrogate pair). At 2 days post-intervention, 2 attrition in the SPIRIT group and 1 attrition in the Comparison group
Measure: Number; unit: Dyads
Arm/Group | SPIRIT-Dementia | Usual Care
Number analyzed (Participants) | 9 | 10
Dyads
  Congruent at Baseline | 1 | 5
  Incongruent at Baseline | 8 | 5
  Congruent at two (2) days post-intervention: number analyzed (Participants) | 7 | 9
  Congruent at two (2) days post-intervention | 1 | 4
  Incongruent at wo (2) days post-intervention: number analyzed (Participants) | 7 | 9
  Incongruent at wo (2) days post-intervention | 6 | 5

2. Primary Outcome: Patient's Decisional Conflict Scale (DCS) Score
Description: Patient decisional conflict will be measured using the 13-item Decisional Conflict Scale (DCS), a validated measure in the context of end-of-life decision making. Participants indicate their level of agreement with statements about their plans for their future medical care by selecting (1) Strongly Agree, (2) Agree, (3) Neither Agree nor Disagree, (4) Disagree, or (5) Strongly Disagree. The total score ranges from 13 - 65 with higher scores indicating greater difficulty in weighing benefits and burdens of life-sustaining treatments and decision making.
Time Frame: Baseline, 2 Days Post-intervention
Population: This analysis includes participants (patients) who completed the indicated study visit. Two participants (patients) in the SPIRIT group and one participant (patient) in the Comparison group did not complete the 2-day post-intervention follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SPIRIT Dementia - Patients: Patients at clinics that have been randomized to the SPIRIT arm will be given the option to participate in the intervention.
  Patients and their surrogates randomized to this study arm will receive the SPIRIT-dementia intervention.
- Comparison Usual Care - Patients: Patients at clinics that have been randomized to the control arm will be given the option to participate as a study control. Patients and surrogates randomized to this study arm will receive the standard information about advance directives that is provided at the time of diagnosis.
Arm/Group | SPIRIT Dementia - Patients | Comparison Usual Care - Patients
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 14.11 (1.62) | 16.00 (2.49)
  Two (2) Days Post-Intervention: number analyzed (Participants) | 7 | 9
  Two (2) Days Post-Intervention | 15.29 (2.21) | 16.67 (3.84)

3. Primary Outcome: Surrogate's Decision Making Confidence (DMC) Scale Score
Description: Surrogate decision-making confidence will be measured using the 5-item Decision Making Confidence (DMC) scale. Surrogates indicate how confident they are about making medical decisions if the patient becomes unable to make their own decisions by their level of agreement with statements along a scale of (0) "Not confident at all" to (5) "Very confident". Total scores range from 0 - 20, with higher scores indicating greater confidence.
Time Frame: Baseline, 2 Days Post-intervention
Population: This analysis includes participants who completed study visits. There were two attrition (surrogates) in the SPIRIT group and one (surrogate) attrition in the Comparison group At 2 days post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SPIRIT Dementia - Surrogates: Surrogates of patients at clinics that have been randomized to the SPIRIT arm will be given the option to participate in the intervention.
  Patients and their surrogates randomized to this study arm will receive the SPIRIT-dementia intervention.
- Comparison Usual Care - Surrogates: Surrogates of patients at clinics that have been randomized to the control arm will be given the option to participate as a study control. Patients and surrogates randomized to this study arm will receive the standard information about advance directives that are provided at the time of diagnosis.
Arm/Group | SPIRIT Dementia - Surrogates | Comparison Usual Care - Surrogates
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 18.44 (1.42) | 17.00 (6.01)
  Two (2) Days Post-Intervention: number analyzed (Participants) | 7 | 9
  Two (2) Days Post-Intervention | 17.57 (4.79) | 18.67 (1.94)

4. Secondary Outcome: Care Decisions (Withdrawal From Dialysis, DNR, Hospice Enrollment)
Description: The proportion of decisions (participants who withdrew from dialysis, Do not resuscitate (DNR), or chose hospice enrollment) will be compared between study arms.
Time Frame: 6 and 12 Months Post-intervention
Population: At both 6 and 12 months post-intervention, 2 attrition in the SPIRIT group and 2 attrition in the Comparison group
Measure: Count of Participants; unit: Participants
Groups:
- SPIRIT Dementia - Patients: Patients at clinics that have been randomized to the SPIRIT arm will be given the option to participate in the intervention.
  Patients and their surrogates randomized to this study arm will receive the SPIRIT-dementia intervention.
  SPIRIT-Dementia: The interventionist will begin the SPIRIT-dementia session by assessing the patient's and surrogate's cognitive, emotional, and spiritual/religious representations of the patient's illness, prognosis, and end-of-life care. Individualized information will be provided about the effectiveness of life-sustaining treatment for people with end-organ failure, and the patient will examine their values about life-sustaining treatment at the end of life. The interventionist will help the surrogate prepare for end-of-life decision-making and for the emotional burden of decision-making. A Goals-of-Care document will be completed at the end of the session. The delivery of SPIRIT-dementia incorporates "enhanced consent techniques," such as reducing information load by proceeding in manageable segments, offering repetition of material, an opportunity for rehearsal, and using targeted questioning to verify adequate comprehension prior to eliciting preferences for goals of care.
- Comparison Usual Care - Patients: Patients and surrogates randomized to this study arm will receive the standard information about advance directives that are provided at the time of diagnosis.
  Usual Care: As required by the Centers for Medicare and Medicaid Services (CMS) written information on advance directives is provided to a patient on the first day of dialysis, and a social worker reviews this information with patients and encourages them to complete an advance directive.
Arm/Group | SPIRIT Dementia - Patients | Comparison Usual Care - Patients
Number analyzed (Participants) | 9 | 10
Participants
  6 months post-intervention: Participants who withdrew from dialysis: number analyzed (Participants) | 7 | 8
  6 months post-intervention: Participants who withdrew from dialysis | 0 | 0
  6 months post-intervention: Participants who chose Do Not Resuscitate (DNR): number analyzed (Participants) | 7 | 8
  6 months post-intervention: Participants who chose Do Not Resuscitate (DNR) | 0 | 0
  6 months post-intervention: Participants who chose Hospice enrollment: number analyzed (Participants) | 7 | 8
  6 months post-intervention: Participants who chose Hospice enrollment | 0 | 0
  12 months post-intervention: Participants who withdrew from dialysis: number analyzed (Participants) | 7 | 8
  12 months post-intervention: Participants who withdrew from dialysis | 0 | 1
  12 months post-intervention Participants who chose Do Not Resuscitate (DNR): number analyzed (Participants) | 7 | 8
  12 months post-intervention Participants who chose Do Not Resuscitate (DNR) | 0 | 1
  12 months post-intervention: Participants who chose Hospice enrollment: number analyzed (Participants) | 7 | 8
  12 months post-intervention: Participants who chose Hospice enrollment | 0 | 0

5. Secondary Outcome: Surrogate's Anxiety-Score Using the Hospital Anxiety and Depression Scale (HADS) Score
Description: Surrogate post-bereavement anxiety and depressive symptoms will be measured with the Hospital Anxiety and Depression Scale (HADS). Surrogates indicate their level of agreement with statements by selecting responses rated from 0 (the problem in the statement is not an issue) to 3 (the problem in the statement is a very big issue). The separate anxiety and depression subscale scores range from 0 to 21 with higher scores indicating greater symptom severity. A score of 0-7 indicates "normal", 8-10 indicates "borderline abnormal", and 11-21 indicates "abnormal" levels of anxiety or depression.
Time Frame: Baseline, 1 Month after the Patient's Death
Population: The surrogate in the SPIRIT group did not complete the post-bereavement assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPIRIT Dementia - Surrogates | Comparison Usual Care - Surrogates
Number analyzed (Participants) | 1 | 2
score on a scale
  Anxiety at Baseline | 2.00 (NA) — Unable to provide standard deviation (SD) on the score of only one (1) participant. | 4.00 (0.00)
  Anxiety - 1 Month after patient' death: number analyzed (Participants) | 0 | 2
  Anxiety - 1 Month after patient' death |  | 7.50 (0.71)

6. Secondary Outcome: Surrogate's Depression-Score by Using the Hospital Anxiety and Depression Scale (HADS) Score
Description: as for outcome 5
Time Frame: Baseline, 1 Month after the Patient's Death
Population: The surrogate in the SPIRIT group did not complete the post-bereavement assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPIRIT Dementia - Surrogates | Comparison Usual Care - Surrogates
Number analyzed (Participants) | 1 | 2
score on a scale
  Depression at Baseline | 7.00 (NA) — Unable to provide standard deviation (SD) on the score of only one (1) participant. | 7.00 (4.24)
  Depression - 1 Month after patient' death: number analyzed (Participants) | 0 | 2
  Depression - 1 Month after patient' death |  | 9.50 (2.12)

ADVERSE EVENTS:
Time Frame: Up to six months after enrollment. Due to the population being examined and the nature of this study, deaths in the patient population are not considered adverse events.
Description: Only adverse events related to the intervention, such as emotional distress, were documented during the intervention session. Due to the population being examined and the nature of this study, deaths are not considered an adverse event in this population, however, known deaths occurring up to the 6-month assessment were documented.
Groups:
- SPIRIT-Dementia- Patients: Patients and their surrogates randomized to this study arm will receive the SPIRIT-dementia intervention.
  SPIRIT-Dementia: The interventionist will begin the SPIRIT-dementia session by assessing the patient's and surrogate's cognitive, emotional, and spiritual/religious representations of the patient's illness, prognosis, and end-of-life care. Individualized information will be provided about the effectiveness of life-sustaining treatment for people with end-organ failure, and the patient will examine their values about life-sustaining treatment at the end of life. The interventionist will help the surrogate prepare for end-of-life decision-making and for the emotional burden of decision-making. A Goals-of-Care document will be completed at the end of the session. The delivery of SPIRIT-dementia incorporates "enhanced consent techniques," such as reducing information load by proceeding in manageable segments, offering repetition of material, opportunity for rehearsal, and using targeted questioning to verify adequate comprehension prior to eliciting preferences for goals of care.
- SPIRIT-Dementia- Surrogates: Surrogates of patients randomized to this study arm will receive the SPIRIT-dementia intervention.
  SPIRIT-Dementia: The interventionist will begin the SPIRIT-dementia session by assessing the patient's and surrogate's cognitive, emotional, and spiritual/religious representations of the patient's illness, prognosis, and end-of-life care. Individualized information will be provided about the effectiveness of life-sustaining treatment for people with end-organ failure, and the patient will examine their values about life-sustaining treatment at the end of life. The interventionist will help the surrogate prepare for end-of-life decision-making and for the emotional burden of decision-making. A Goals-of-Care document will be completed at the end of the session. The delivery of SPIRIT-dementia incorporates "enhanced consent techniques," such as reducing information load by proceeding in manageable segments, offering repetition of material, opportunity for rehearsal, and using targeted questioning to verify adequate comprehension prior to eliciting preferences for goals of care.
- Usual Care - Surrogates: Patients and surrogates randomized to this study arm will receive the standard information about advance directives that are provided at the time of diagnosis.
  Usual Care: As required by the Centers for Medicare and Medicaid Services (CMS) written information on advance directives is provided to a patient on the first day of dialysis, and a social worker reviews this information with patients and encourages them to complete an advance directive.
Arm/Group | SPIRIT-Dementia- Patients | SPIRIT-Dementia- Surrogates | Usual Care - Patients | Usual Care - Surrogates
All-Cause Mortality (participants affected / at risk) | 1/9 | 1/9 | 1/10 | 1/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT04108000/Prot_SAP_001.pdf
  • Informed Consent Form (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT04108000/ICF_000.pdf